CLINICAL TRIAL: NCT03363178
Title: A Single-arm, Open-label, Single-center, Phase 1 Study to Investigate the Safety and Efficacy of GC3107 (BCG Vaccine) After Intradermal Administration in Healthy Adults
Brief Title: Study to Investigate the Safety and Efficacy of GC3107 (BCG Vaccine) in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GC3107_P1
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GC3107 (Experimental): BCG Vaccine, 0.1mL
  Interventions: Biological: GC3107

INTERVENTIONS:
Biological: GC3107 — BCG Vaccine, 0.1mL

SUMMARY:
Healthy adults will be once administered GC3107(BCG Vaccine) Intradermally.

DETAILED DESCRIPTION:
Healthy adults will be once administered GC3107(BCG Vaccine) Intradermally. Tuberculin Skin Test(TST) will be conducted after 84+7 days after IP injection and TST result will be read in 48~72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19-64 years old
* Informed consent form has been signed and dated
* Able to comply with the requirements of the study
* Female subjects who have negative results in Urine hCG test at screening, or menopausal women.

Exclusion Criteria:

* Subjects who have positive results(;induration diameter over 5mm) in Tuberculin Skin Test(TST) at screening
* Subjects who shown abnormal results(including inactive tuberculosis) on Chest X-ray at screening
* Subjects who received a vaccination(including live vaccine) within 28 days before enrollment
* Subjects who are on antituberculosis drugs
* Immunocompromised subjects with immunodeficiency disease or subjects receiving immunosuppressive or immunomodulating therapy
* Subjects with severe chronic disease who are considered by investigator to be ineligible for the study
* Pregant or lactating women

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | for 7 days from Day0/during study period
  Solicited/Unsolicited Adverse Event

SECONDARY OUTCOMES:
Whether the maximum Induration diameter greater than 5mm after TST. | Day0+84days
  Induration diameter measured in the direction perpendicular to the arm.
Whether the maximum Erythema/Redness diameter greater than 5mm after TST. | Day0+84days
  Erythema/Redness diameter measured in the direction perpendicular to the arm.
Maximum diameter of Induration after TST. | Day0+84days
  Induration diameter measured in the direction perpendicular to the arm.
Maximum diameter of Erythema/Redness after TST. | Day0+84days
  Erythema/Redness diameter measured in the direction perpendicular to the arm.
Maximum diameter variation of Induration after TST. | Day0+84days
  Induration diameter measured in the direction perpendicular to the arm.
Maximum diameter variation of Erythema/Redness after TST. | Day0+84days
  Erythema/Redness diameter measured in the direction perpendicular to the arm.

CONTACTS AND LOCATIONS:
Overall Officials: Woo Joo Kim, M.D, Ph.D, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No